CLINICAL TRIAL: NCT02630992
Title: Reduced Clavulanate Formulation of Amoxicillin-Clavulanate in Children 6-23 Months With Acute Otitis Media
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nader Shaikh (Other)
Responsible Party: Sponsor-Investigator, Nader Shaikh, Associate Professor of Pediatrics, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRO15080192
Record Dates: First submitted 2015-12-11; First posted 2015-12-15 (Estimated); Results first posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Acute Otitis Media
Keywords: ear infections; antibiotics; antibiotic resistance; pediatrics; infants; children; amoxicillin-clavulanate
MeSH Terms: conditions — Otitis Media; Otitis | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- amoxicillin-clavulanate potassium (Experimental): amoxicillin-clavulanate potassium (600 mg/221.5 mg/5 mL; 28:1) administered prior to February 25, 2016 at 90/3.2 mg/kg/day in two divided doses for 10 days; oral, liquid (formulation 1) or administered as of February 25, 2016 at 80/2.85 mg/kg/day in two divided doses for 10 days; oral, liquid (formulation 2)
  Interventions: Drug: Amoxicillin-Clavulanate potassium

INTERVENTIONS:
Drug: Amoxicillin-Clavulanate potassium
  Other Names: Augmentin

SUMMARY:
To evaluate the safety profile of amoxicillin-clavulanate potassium containing a reduced concentration of clavulanate potassium, 600 mg/21.5 mg/5 mL (a ratio of 28:1), administered at 90/3.2 mg/kg/day (formulation 1) or at 80/2.85 mg/kg/day (formulation 2) in two divided doses for 10 days. Investigators will focus on the proportion of subjects who develop protocol-defined diarrhea and proportion who develop diaper dermatitis that occasions the prescription of antifungal medication.

DETAILED DESCRIPTION:
Amoxicillin-clavulanate potassium has been shown to be efficacious in eradicating causative pathogens in acute otitis media (AOM) with resulting high clinical cure rates at end-of-treatment (85%). However, relatively high rates (~25%) of clinically significant diarrhea have been reported, the occurrence of which has been directly related to the clavulanate potassium component of the drug combination. A reduced concentration of clavulanate potassium in the drug formulation would be expected to have an improved safety profile regarding the occurrence of diarrhea. This study will examine whether the concentration of the clavulanate potassium component of amoxicillin-clavulanate potassium could be reduced in the treatment of children 6 months through 23 months of age diagnosed with AOM using stringent criteria. A total of 75 participants (n=75) with AOM will receive amoxicillin-clavulanate potassium (600 mg/21.5 mg/5 mL; 28:1) administered at 90/3.2 mg/kg/day (formulation 1) or at 80/2.85 mg/kg/day (formulation 2) in two divided doses for 10 days.

The primary outcome measure will be rates of clinically significant diarrhea and diaper dermatitis. These rates will be compared with the rate observed in our previous studies of AOM in children who received amoxicillin-clavulanate potassium (600 mg/42.9 mg/5 mL; 14:1) administered at 90/6.4 mg/kg/day in two divided doses for 10 days.

A subset of this group will have pharmacokinetic studies performed. Each participant that agrees will have a single blood draw (n=50). Investigators will analyze amoxicillin and clavulanate potassium in the blood samples using validated methods.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 6 to 23 months
* Evidence of AOM
* Recent (within 48 hours) onset of signs and symptoms.
* Middle ear effusion evidenced by the presence of at least 2 of the following: decreased or absent mobility of the tympanic membrane (TM), yellow of white discoloration of the TM, and/or opacification of the TM
* Acute inflammation evidenced by one of the following: 1+ bulging of the TM with either intense erythema or otalgia or 2+ or 3+ bulging of the TM

Exclusion Criteria:

* Toxic appearance (capillary refill >3 seconds, systolic blood pressure <60 mm Hg)
* Inpatient hospitalization
* Clinical or anatomical characteristics that might obscure response to treatment (e.g., tympanostomy tubes in place, cleft palate, Down syndrome)
* Sensorineural hearing loss (unilateral or bilateral)
* Allergy to amoxicillin or amoxicillin clavulanate
* Recent treatment of AOM within the last 14 days

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nader Shaikh, MD, MPH, Principal Investigator — University of Pittsburgh School of Medicine; Children's Hospital of Pittsburgh of UPMC
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoberman A, Paradise JL, Rockette HE, Jeong JH, Kearney DH, Bhatnagar S, Shope TR, Muniz G, Martin JM, Kurs-Lasky M, Haralam M, Pope MA, Nagg JP, Zhao W, Miah MK, Beumer J, Venkataramanan R, Shaikh N. Reduced-Concentration Clavulanate for Young Children with Acute Otitis Media. Antimicrob Agents Chemother. 2017 Jun 27;61(7):e00238-17. doi: 10.1128/AAC.00238-17. Print 2017 Jul. PMID 28438923

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amoxicillin-clavulanate Potassium
Started | 112
Completed | 99
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Amoxicillin-clavulanate Potassium
Number analyzed (Participants) | 112
Age, Customized [Count of Participants; unit: Participants]
  6-11 months | 59
  12-23 months | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was reported by the children's parents.
  Participants
    Hispanic or Latino | 12
    Not Hispanic or Latino | 99
    Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race was reported by the children's parents.
  Participants
    American Indian or Alaska Native | 0
    Asian | 5
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 74
    White | 17
    More than one race | 13
    Unknown or Not Reported | 3
Maternal Education [Count of Participants; unit: Participants]
  Below high school graduate | 7
  High school graduate or equivalent | 80
  College graduate | 24
  Unknown | 1
Type of Health Insurance [Count of Participants; unit: Participants] — Type of health insurance relates to the child's insurance.
  Participants
    Private | 34
    Public | 78
Exposure to Other Children [Count of Participants; unit: Participants] — Exposed to other children is defined as exposure to at least 3 children for at least 10 hours per week.
  Participants
    No | 47
    Yes | 65
Acute Otitis Media Severity of Symptoms (AOM-SOS) Score [Count of Participants; unit: Participants] — The AOM-SOS scale measures five discrete items: tugging of ears, crying, irritability, difficulty sleeping, and fever. Parents are asked to rate these symptoms in comparison with the child's usual state, as "none," "a little," or "a lot," with corresponding scores of 0, 1, and 2. Thus, total scores range from 0 to 10, with higher scores indicating greater severity of symptoms.
  Participants
    3-5 | 40
    6-8 | 50
    9-10 | 22
Mean AOM-SOS Score [Mean (Standard Deviation); unit: AOM-SOS score] — The AOM-SOS scale measures five discrete items: tugging of ears, crying, irritability, difficulty sleeping, and fever. Parents are asked to rate these symptoms in comparison with the child's usual state, as "none," "a little," or "a lot," with corresponding scores of 0, 1, and 2. Thus, total scores range from 0 to 10, with higher scores indicating greater severity of symptoms.
  AOM-SOS score | 6.4 (2.0)
Laterality of Acute Otitis Media (AOM) [Count of Participants; unit: Participants]
  Unilateral | 65
  Bilateral | 47
Degree of Tympanic Membrane (TM) Bulging [Count of Participants; unit: Participants] — If a child has unilateral AOM, the degree of bulging reflects the degree of bulging in the ear with AOM. If a child has bilateral AOM, the degree of bulging reflects the degree of bulging in the ear with the greater level of bulging,
  Participants
    Slight | 9
    Moderate or marked | 103

OUTCOME MEASURES:

1. Primary Outcome: The Distribution of Participants Receiving Formulation 1 for Whom Protocol-Defined Diarrhea (PDD) Was Reported and Associated With Study Product
Description: Participants receiving formulation 1 were administered amoxicillin-clavulanate potassium containing a reduced concentration of clavulanate potassium, 600 mg/21.5 mg/5 mL (a ratio of 28:1), administered at 90/3.2 mg/kg/day in two divided doses for 10 days.
  Protocol-defined diarrhea is defined as the occurrence of three or more watery stools in 1 day or two watery stools daily for 2 consecutive days and is limited to events associated with study product.
Time Frame: Day 1 of administration of amoxicillin-clavulanate until day 12.
Population: The number of participants is equal to the number of children receiving formulation 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin-clavulanate Potassium
Number analyzed (Participants) | 40
Participants
  PDD reported | 10
  PDD not reported | 30

2. Primary Outcome: The Distribution of Participants Receiving Formulation 2 for Whom Protocol-Defined Diarrhea (PDD) Was Reported and Associated With Study Product
Description: Participants receiving formulation 2 were administered amoxicillin-clavulanate potassium containing a reduced concentration of clavulanate potassium, 600 mg/21.5 mg/5 mL (a ratio of 28:1), administered at 80/2.85 mg/kg/day in two divided doses for 10 days.
  Protocol-defined diarrhea is defined as the occurrence of three or more watery stools in 1 day or two watery stools daily for 2 consecutive days and is limited to events associated with study product.
Time Frame: Day 1 of administration of amoxicillin-clavulanate until day 12.
Population: The number of participants is equal to the number of children receiving formulation 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin-clavulanate Potassium
Number analyzed (Participants) | 72
Participants
  PDD reported | 12
  PDD not reported | 60

3. Primary Outcome: The Distribution of Participants Receiving Formulation 1 for Whom Diaper Dermatitis Was Reported and Associated With Study Product
Description: Participants receiving formulation 1 were administered amoxicillin-clavulanate potassium containing a reduced concentration of clavulanate potassium, 600 mg/21.5 mg/5 mL (a ratio of 28:1), administered at 90/3.2 mg/kg/day in two divided doses for 10 days.
  Diaper dermatitis is defined as dermatitis in the diaper area calling for prescription of a topical antifungal agent and is limited to events associated with study product.
Time Frame: Day 1 of administration of amoxicillin-clavulanate until day 12.
Population: The number of participants is equal to the number of children receiving formulation 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin-clavulanate Potassium
Number analyzed (Participants) | 40
Participants
  Diaper dermatitis reported | 10
  Diaper dermatitis not reported | 30

4. Primary Outcome: The Distribution of Participants Receiving Formulation 2 for Whom Diaper Dermatitis Was Reported and Associated With Study Product
Description: Participants receiving formulation 2 were administered amoxicillin-clavulanate potassium containing a reduced concentration of clavulanate potassium, 600 mg/21.5 mg/5 mL (a ratio of 28:1), administered at 80/2.85 mg/kg/day in two divided doses for 10 days.
  Diaper dermatitis is defined as dermatitis in the diaper area calling for prescription of a topical antifungal agent and is limited to events associated with study product..
Time Frame: Day 1 of administration of amoxicillin-clavulanate until day 12.
Population: The number of participants is equal to the number of children receiving formulation 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin-clavulanate Potassium
Number analyzed (Participants) | 72
Participants
  Diaper dermatitis reported | 15
  Diaper dermatitis not reported | 57

5. Secondary Outcome: The Distribution of Participants Receiving Formulation 1 Categorized as Treatment Failure (TF) at or Before the End-of-Treatment Visit
Description: Participants receiving formulation 1 were administered amoxicillin-clavulanate potassium containing a reduced concentration of clavulanate potassium, 600 mg/21.5 mg/5 mL (a ratio of 28:1), administered at 90/3.2 mg/kg/day in two divided doses for 10 days.
  Treatment failure is defined as substantial persistence or worsening of symptoms specifically attributable to AOM or of otoscopic signs of acute inflammation (bulging of the TM or intense erythema) after 72 hours from the initial AOM, such that additional antimicrobial therapy is deemed advisable. Clinical success is defined as complete or substantial resolution of symptoms specifically attributable to AOM for 48 hours and of otoscopic signs of acute inflammation (bulging of the TM or intense erythema), with or without persistence of middle-ear effusion, such that no additional antibiotic therapy is deemed advisable.
Time Frame: From 72 hours after the initial AOM until the end-of-treatment visit. The mean day for this visit was 14.9.
Population: The number of participants is equal to the number of children receiving formulation 1 who had an end-of-treatment assessment at or before the day 12 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin-clavulanate Potassium
Number analyzed (Participants) | 35
Participants
  Treatment failure | 4
  Clinical success | 31

6. Secondary Outcome: The Distribution of Participants Receiving Formulation 2 Categorized as Treatment Failure (TF) at or Before the End-of-Treatment Visit
Description: Participants receiving formulation 2 were administered amoxicillin-clavulanate potassium containing a reduced concentration of clavulanate potassium, 600 mg/21.5 mg/5 mL (a ratio of 28:1), administered at 80/2.85 mg/kg/day in two divided doses for 10 days.
  Treatment failure is defined as substantial persistence or worsening of symptoms specifically attributable to AOM or of otoscopic signs of acute inflammation (bulging of the TM or intense erythema) after 72 hours from the initial AOM, such that additional antimicrobial therapy is deemed advisable. Clinical success is defined as complete or substantial resolution of symptoms specifically attributable to AOM for 48 hours and of otoscopic signs of acute inflammation (bulging of the TM or intense erythema), with or without persistence of middle-ear effusion, such that no additional antibiotic therapy is deemed advisable.
Time Frame: From 72 hours after the initial AOM until the end-of-treatment visit. The mean day for this visit was 13.9.
Population: The number of participants is equal to the number of children receiving formulation 2 who had an end-of-treatment assessment at or before the day 12 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin-clavulanate Potassium
Number analyzed (Participants) | 64
Participants
  Treatment failure | 8
  Clinical success | 56

7. Secondary Outcome: The Distribution of Participants Receiving Formulation 1 Demonstrating Resolution of Acute Otitis Media (AOM) and Substantial Improvement of Symptoms That Would Allow Discontinuing Therapy at the Day 7 Visit
Description: Participants receiving formulation 1 were administered amoxicillin-clavulanate potassium containing a reduced concentration of clavulanate potassium, 600 mg/21.5 mg/5 mL (a ratio of 28:1), administered at 90/3.2 mg/kg/day in two divided doses for 10 days.
  An assessment of participants was conducted at the day 7 visit using the AOM-SOS scale.
  The AOM-SOS scale measures five discrete items: tugging of ears, crying, irritability, difficulty sleeping, and fever. Parents are asked to rate these symptoms in comparison with the child's usual state, as "none," "a little," or "a lot," with corresponding scores of 0, 1, and 2. Thus, total scores range from 0 to 10, with higher scores indicating greater severity of symptoms.
Time Frame: Day 1 of administration of amoxicillin-clavulanate until the day 7 visit. The mean day for this visit was 7.5.
Population: The number of participants is equal to the number of children receiving formulation 1 who had a day 7 assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin-clavulanate Potassium
Number analyzed (Participants) | 34
Participants
  Resolution of AOM and improvement of symptoms | 23
  No resolution of AOM or no improvement of symptoms | 11

8. Secondary Outcome: The Distribution of Participants Receiving Formulation 2 Demonstrating Resolution of Acute Otitis Media (AOM) and Substantial Improvement of Symptoms That Would Allow Discontinuing Therapy at the Day 7 Visit
Description: Participants receiving formulation 2 were administered amoxicillin-clavulanate potassium containing a reduced concentration of clavulanate potassium, 600 mg/21.5 mg/5 mL (a ratio of 28:1), administered at 80/2.85 mg/kg/day in two divided doses for 10 days.
  An assessment of participants was conducted at the day 7 visit using the AOM-SOS scale.
  The AOM-SOS scale measures five discrete items: tugging of ears, crying, irritability, difficulty sleeping, and fever. Parents are asked to rate these symptoms in comparison with the child's usual state, as "none," "a little," or "a lot," with corresponding scores of 0, 1, and 2. Thus, total scores range from 0 to 10, with higher scores indicating greater severity of symptoms.
Time Frame: Day 1 of administration of amoxicillin-clavulanate until the day 7 visit. The mean day for this visit was 7.6.
Population: The number of participants is equal to the number of children receiving formulation 2 who had a day 7 assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin-clavulanate Potassium
Number analyzed (Participants) | 62
Participants
  Resolution of AOM and improvement of symptoms | 31
  No resolution of AOM or no improvement of symptoms | 31

9. Secondary Outcome: The Mean Score Representing the Parent or Guardian's Level of Satisfaction With Therapy for Participants Receiving Formulation 1
Description: Participants receiving formulation 1 were administered amoxicillin-clavulanate potassium containing a reduced concentration of clavulanate potassium, 600 mg/21.5 mg/5 mL (a ratio of 28:1), administered at 90/3.2 mg/kg/day in two divided doses for 10 days.
  The parent or guardian will answer a questionnaire regarding their satisfaction with the therapy their child received. The responses 'very dissatisfied', 'somewhat dissatisfied', 'neither satisfied nor dissatisfied', 'somewhat satisfied' and 'very satisfied' correspond to scores of 1, 2, 3, 4, and 5, respectively.
Time Frame: The end-of-treatment visit. The mean day for this visit was 14.9.
Population: The number of participants is equal to the number of children receiving formulation 1 whose parent or guardian completed a level of satisfaction questionnaire at the end-of-treatment visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Amoxicillin-clavulanate Potassium
Number analyzed (Participants) | 35
units on a scale | 4.69 (0.72)

10. Secondary Outcome: The Mean Score Representing the Parent or Guardian's Level of Satisfaction With Therapy for Participants Receiving Formulation 2
Description: Participants receiving formulation 2 were administered amoxicillin-clavulanate potassium containing a reduced concentration of clavulanate potassium, 600 mg/21.5 mg/5 mL (a ratio of 28:1), administered at 80/2.85 mg/kg/day in two divided doses for 10 days.
  The parent or guardian will answer a questionnaire regarding their satisfaction with the therapy their child received. The responses 'very dissatisfied', 'somewhat dissatisfied', 'neither satisfied nor dissatisfied', 'somewhat satisfied' and 'very satisfied' correspond to scores of 1, 2, 3, 4, and 5, respectively.
Time Frame: The end-of-treatment visit. The mean day for this visit was 13.9.
Population: The number of participants is equal to the number of children receiving formulation 2 whose parent or guardian completed a level of satisfaction questionnaire at the end-of-treatment visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Amoxicillin-clavulanate Potassium
Number analyzed (Participants) | 64
units on a scale | 4.75 (0.76)

11. Secondary Outcome: Distribution of Population Plasma Concentration of Amoxicillin According to Time For Participants Receiving Formulation 1
Description: Participants receiving formulation 1 were administered amoxicillin-clavulanate potassium containing a reduced concentration of clavulanate potassium, 600 mg/21.5 mg/5 mL (a ratio of 28:1), administered at 90/3.2 mg/kg/day in two divided doses for 10 days.
  Plasma concentration of amoxicillin 45 mg/kg/dose was measured.
  Data points up to 4 hours with a standard deviation of 0 indicate that the assessment was available for only one child.
Time Frame: From administration of a single dose of amoxicillin-clavulanate until approximately 4 hours after.
Population: The participants are the children receiving formulation 1 whose parent or guardian agreed to a single blood draw after administration of a single dose of amoxicillin-clavulanate and who had an ensuing measure of plasma concentration.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/ml)
Arm/Group | Amoxicillin-clavulanate Potassium
Number analyzed (Participants) | 15
micrograms per milliliter (mcg/ml)
  0.5 hours (approximate): number analyzed (Participants) | 3
  0.5 hours (approximate) | 14.36 (10.07)
  1.5 hours (approximate): number analyzed (Participants) | 1
  1.5 hours (approximate) | 15.3 (0)
  2.0 hours (approximate): number analyzed (Participants) | 4
  2.0 hours (approximate) | 11.42 (5.00)
  3.0 hours (approximate): number analyzed (Participants) | 1
  3.0 hours (approximate) | 8.07 (0)
  3.5 hours (approximate): number analyzed (Participants) | 1
  3.5 hours (approximate) | 9.78 (0)
  4.0 hours (approximate): number analyzed (Participants) | 5
  4.0 hours (approximate) | 7.39 (8.33)

12. Secondary Outcome: Distribution of Population Plasma Concentration of Amoxicillin According to Time For Participants Receiving Formulation 2
Description: Participants treated with formulation 2 were administered amoxicillin-clavulanate potassium containing a reduced concentration of clavulanate potassium, 600 mg/21.5 mg/5 mL (a ratio of 28:1), administered at 80/2.85 mg/kg/day in two divided doses for 10 days.
  Plasma concentration of amoxicillin 40 mg/kg/dose was measured.
  Data points up to 4 hours with a standard deviation of 0 indicate that the assessment was available for only one child.
Time Frame: From administration of a single dose of amoxicillin-clavulanate until approximately 4 hours after.
Population: The participants are the children receiving formulation 2 whose parent or guardian agreed to a single blood draw after administration of a single dose of amoxicillin-clavulanate and who had an ensuing measure of plasma concentration.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/ml)
Arm/Group | Amoxicillin-clavulanate Potassium
Number analyzed (Participants) | 24
micrograms per milliliter (mcg/ml)
  0.5 hours (approximate): number analyzed (Participants) | 3
  0.5 hours (approximate) | 8.63 (3.89)
  1.5 hours (approximate): number analyzed (Participants) | 2
  1.5 hours (approximate) | 7.49 (1.59)
  2.0 hours (approximate): number analyzed (Participants) | 4
  2.0 hours (approximate) | 7.76 (6.56)
  2.5 hours (approximate): number analyzed (Participants) | 7
  2.5 hours (approximate) | 10.22 (7.18)
  3.0 hours (approximate): number analyzed (Participants) | 2
  3.0 hours (approximate) | 13.00 (0.50)
  3.5 hours (approximate): number analyzed (Participants) | 2
  3.5 hours (approximate) | 10.36 (1.94)
  4.0 hours (approximate): number analyzed (Participants) | 4
  4.0 hours (approximate) | 8.52 (4.54)

13. Secondary Outcome: Distribution of Population Plasma Concentration of Clavulanate According to Time For Participants Receiving Formulation 1
Description: Participants receiving formulation 1 were administered amoxicillin-clavulanate potassium containing a reduced concentration of clavulanate potassium, 600 mg/21.5 mg/5 mL (a ratio of 28:1), administered at 90/3.2 mg/kg/day in two divided doses for 10 days.
  Plasma concentration of clavulanate 1.6 mg/kg/dose was measured.
  Data points up to 4 hours with a standard deviation of 0 indicate that the assessment was available for only one child.
Time Frame: From administration of a single dose of amoxicillin-clavulanate until approximately 4 hours after.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/ml)
Arm/Group | Amoxicillin-clavulanate Potassium
Number analyzed (Participants) | 15
nanograms per milliliter (ng/ml)
  0.5 hours (approximate): number analyzed (Participants) | 3
  0.5 hours (approximate) | 1047.67 (419.90)
  1.5 hours (approximate): number analyzed (Participants) | 1
  1.5 hours (approximate) | 2050 (0)
  2.0 hours (approximate): number analyzed (Participants) | 4
  2.0 hours (approximate) | 730.50 (442.93)
  3.0 hours (approximate): number analyzed (Participants) | 1
  3.0 hours (approximate) | 338 (0)
  3.5 hours (approximate): number analyzed (Participants) | 1
  3.5 hours (approximate) | 842 (0)
  4.0 hours (approximate): number analyzed (Participants) | 5
  4.0 hours (approximate) | 313.80 (146.91)

14. Secondary Outcome: Distribution of Population Plasma Concentration of Clavulanate According to Time For Participants Receiving Formulation 2
Description: Participants receiving formulation 2 were administered amoxicillin-clavulanate potassium containing a reduced concentration of clavulanate potassium, 600 mg/21.5 mg/5 mL (a ratio of 28:1), administered at 80/2.85 mg/kg/day in two divided doses for 10 days.
  Plasma concentration of clavulanate 1.425 mg/kg/dose was measured.
  Data points up to 4 hours with a standard deviation of 0 indicate that the assessment was available for only one child.
Time Frame: From administration of a single dose of amoxicillin-clavulanate until approximately 4 hours after.
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/ml)
Arm/Group | Amoxicillin-clavulanate Potassium
Number analyzed (Participants) | 23
nanograms per milliliter (ng/ml)
  0.5 hours (approximate): number analyzed (Participants) | 3
  0.5 hours (approximate) | 407 (335.47)
  1.5 hours (approximate): number analyzed (Participants) | 2
  1.5 hours (approximate) | 655.50 (20.5)
  2.0 hours (approximate): number analyzed (Participants) | 3
  2.0 hours (approximate) | 1125.33 (418.49)
  2.5 hours (approximate): number analyzed (Participants) | 7
  2.5 hours (approximate) | 660.16 (389.69)
  3.0 hours (approximate): number analyzed (Participants) | 2
  3.0 hours (approximate) | 986.95 (963.05)
  3.5 hours (approximate): number analyzed (Participants) | 2
  3.5 hours (approximate) | 866.00 (534.00)
  4.0 hours (approximate): number analyzed (Participants) | 4
  4.0 hours (approximate) | 555.50 (494.53)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through the end-of-treatment visit. The mean day for this visit was 14.2.
Groups:
- Amoxicillin-clavulanate Potassium: amoxicillin-clavulanate potassium (600 mg/221.5 mg/5 mL; 28:1) administered prior to February 25, 2016 at 90/3.2 mg/kg in two divided doses for 10 days; oral, liquid (formulation 1) or administered as of February 25, 2016 at 80/2.85 mg/kg in two divided doses for 10 days; oral, liquid (formulation 2)
Arm/Group | Amoxicillin-clavulanate Potassium
All-Cause Mortality (participants affected / at risk) | 0/112
Serious Adverse Events (participants affected / at risk) | 0/112
Other Adverse Events (participants affected / at risk) | 38/112
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amoxicillin-clavulanate Potassium (N=112)
Protocol defined diarrhea (Gastrointestinal disorders) | 24 (24) — Protocol defined diarrhea is defined as the occurrence of three or more watery stools in 1 day or two watery stools daily for 2 consecutive days.
Diaper dermatitis (Skin and subcutaneous tissue disorders) | 28 (28) — Diaper dermatitis is defined as dermatitis in the diaper area calling for prescription of a topical antifungal agent.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes